Pokfulam Road, Hong Kong

# Early Socioemotional Intervention for Children with Autism Spectrum Disorder in Hong Kong and Mainland China

NCT number: N/A

Document date: December 7, 2020

Tel: (852) 3917 2375

Fax: (852) 2858 3518

E-mail: dpsychol@hkucc.hku.hk

Web: http://www.hku.hk/psychology



# The University of Hong Kong Department of Psychology

Pokfulam Road, Hong Kong

#### **Research Study on Early Social Skills**

#### Parent/Guardian Consent Form

Dear Parents/Guardians,



We are pleased to inform you about a new research study conducted by our research team led by Prof. Terry Au (Department of Psychology, the University of Hong Kong) and Dr. Lamei Wang (College of Psychology, Shenzhen University) on young children's social skills. This study aims to understand better everyday functioning of young children in China and how to coach parents to support the children's development. We cordially invite you and your child (age 3-6) to participate in this study. We will also invite your child's kindergarten teacher to participate.

In order to better understand their social skills, we hope that your child participate in one-on-one interactive activities with our researcher. The activities will take about an hour. We will also talk to you on the phone for about 1-2 hours about your child's development. You will be asked to complete a set of questionnaires on some basic demographic information and the child's socioemotional and cognitive functioning. Afterwards, we will invite some parents/guardians who are interested in a free parenting program to improve the children's early social skills, which will be conducted by qualified professionals at the Shenzhen University.

Taking part in this study will pose no risk to you and your child. Participation is entirely voluntary, which means that you and your child can withdraw from the research project at any time without any problems. We will explain to your child that they can decide whether to participate and can stop when they wish. All information obtained will remain strictly confidential and will be used for research purposes only. You and your child will not be identified by name in any research reports. Once data collection is completed, all names will be removed from the data records permanently. All records will be destroyed 3 years after publication of the relevant results. If you have any questions about the project, please feel free to contact xxx through phone (xxx). If you want to know more about the rights as a research participant, please contact the Human Research Ethics Committee, the University of Hong Kong (+852 2241-5267) or Human Research Ethics Committee of Health Science Center, Shenzhen University (0755-86930142).

Tel: (852) 3917 2375 Fax: (852) 2858 3518 E-mail: dpsychol@hkucc.hku.hk Web: http://www.hku.hk/psychology

Please complete the reply slip below to indicate whether you would participate and allow your child to participate in this research and return the slip to your child's class teacher by DD/MM/YYYY.

Your help is very much appreciated.

Yours Sincerely,

Prof. Terry Au

Chair Professor

Department of Psychology

The University of Hong Kong

Dr. Lamei Wang

Associate Professor

College of Psychology

Shenzhen University



Pokfulam Road, Hong Kong

## **Research Study on Early Social and Learning Skills**

## **Reply Slip**

| I ** will / will not (** Please circle if appropriate) agree to participate, and give permission to my | |
|---|---|
| child | (child's name),(child's class), to participate in this |
| resear | ch. |
| | I understand that the information obtained from this research can be used for future research and academic publications. However, my and my child's personal data will be kept strictly confidential. |
| | I understand the information stated in the consent form above, and that my and my child's participation in this research is entirely voluntary. |
| | I understand that my child and I have the right to raise any questions during this research and to withdraw from the research at any time without any negative consequences. |
| | Parent Name: Parent Signature: |
| | Parent Contact Number: |
| | Date: |

[HREC Reference Number: EA1811014]



# The University of Hong Kong Department of Psychology

Pokfulam Road, Hong Kong

#### Research Study on Early Social Skills





Dear Principal/Director,

We are pleased to inform you about a new research study conducted by our research team, led by Prof. Terry Au from the Department of Psychology at the University of Hong Kong and Dr. Lamei Wang from the College of Psychology at Shenzhen University, on young children's early social skills. This study aims to understand better young children's social skills and to develop training programs designed for Chinese parents/guardians to help children enhance these important skills. Some parents of students from your institution have signed up to participate in our project; in order better understand the children's social functioning skills, we would also like to invite their teachers to participate in this project.

For children participating in our study, their teachers will be invited to complete a set of questionnaires on the children's socioemotional and cognitive functioning. We will then invite their parents/guardians to join the parenting programs conducted by our research team. Afterwards, the teachers will be asked to re-rate the children's functioning both immediately and 4-month after the parenting program.

The teachers' participation is most important to our research. Taking part in this study will pose no risk to your students, their parents, and teachers. Participation is entirely voluntary, which means that they can choose to withdraw at any time without problems. All information obtained will remain strictly confidential and will be used for research purposes only. Participants will not be identified by name in any research reports. Once data collection is completed, all participating children's and adults' names will be removed from the data records permanently. All records will be destroyed 3 years after publication of the relevant results.

If you have any objection to the teachers' participation in our project, please inform the relevant teachers who has delivered this letter to you. If you want to know more about the rights as a research participant, please contact the Human Research Ethics Committee, the University of Hong Kong (+852 2241-5267) or Human Research Ethics Committee of Health Science Center, Shenzhen University (0755-86930142).

Tel: (852) 3917 2375 Fax: (852) 2858 3518 E-mail: dpsychol@hkucc.hku.hk Web: http://www.hku.hk/psychology

Your support will be most helpful for the success of our research.

Yours Sincerely,

Prof. Terry Au Chair Professor Department of Psychology The University of Hong Kong Dr. Lamei Wang Associate Professor College of Psychology Shenzhen University

# The University of Hong Kong Department of Psychology

Pokfulam Road, Hong Kong

#### Research Study on Early Social Skills

#### **Teacher Consent Form**



Dear Teacher,

We are pleased to inform you about a new research study conducted by our research team, led by Prof. Terry Au from the Department of Psychology at the University of Hong Kong and Dr. Lamei Wang from the College of Psychology at Shenzhen University, on young children's early social skills. This study aims to understand better young children's social skills and to develop training programs designed for Chinese parents/guardians to help children enhance these important skills. In addition to inviting children (age 3-6) and their parents to participate in this study, we would also like to invite you to participate by offering your ideas and observations of the participating children.

During the study, you will be asked to complete a set of questionnaires on the participating child regarding their socioemotional and cognitive functioning. We will then invite their parents/guardians to join the parenting programs conducted by our research team. Afterwards, you will be asked to re-rate the children's functioning both immediately and 4-month after the parenting program. To express our gratitude towards your participation, you will receive RMB100 for each hour of participation and a certificate of appreciation.

Your participation is most important in our research. Taking part in this study will pose no risk to you and the children. Participation is entirely voluntary, which means that you can choose to withdraw at any time without problems. All information obtained will remain strictly confidential and will be used for research purposes only. You will not be identified by name in any research reports. Once data collection is completed, all names will be removed from the data records permanently. All records will be destroyed 3 years after publication of the relevant results. If you have any questions about the project, please feel free to contact xxx through phone (xxx). If you want to know more about the rights as a research participant, please contact the Human Research Ethics Committee at the University of Hong Kong (+852 2241-5267) and the Human Research Ethics Committee of Health Science Center, Shenzhen University (0755-86930142).

Tel: (852) 3917 2375

Fax: (852) 2858 3518

E-mail: dpsychol@hkucc.hku.hk

Web: http://www.hku.hk/psychology

| Please complete the reply slip | below to indicate whether you | would participate | in this resea | ırch |
|---|---|---|---|---|
| and return the slip to our researcher | by DD/MM/YYYY. | | | |

Your help is very much appreciated.

Yours Sincerely,

Prof. Terry Au Chair Professor Department of Psychology The University of Hong Kong Dr. Lamei Wang
Associate Professor
College of Psychology
Shenzhen University

\*\*\*\*\*\*\*\*\*\*\*\*\*\*\*\*\*\*\*\*\*\*



Pokfulam Road, Hong Kong

### **Research Study on Early Social and Learning Skills**

## **Reply Slip**

| I_ | (name) ** wi | 1 / will not (** Please circle if appropriate) agree to |
|---|---|---|
| participa | ate in the research described above | e. |
| | | obtained from this research can be used for future research ver, my personal data will be kept strictly confidential. |
| | understand the information state esearch is entirely voluntary. | d in the consent form above, and that my participation in this |
| | understand that I have the right<br>from the research at any time wit | to raise any questions during this research and to withdraw nout any negative consequences. |
| Teacher | 's name: | Class: |
| Contact number: | | Signature: |
| Date: | | |
| [HREC] | Reference Number: EA1811014 | |

Tel: (852) 3917 2375

Fax: (852) 2858 3518

E-mail: dpsychol@hkucc.hku.hk

Web: http://www.hku.hk/psychology